CLINICAL TRIAL: NCT03710564
Title: A Multicenter, Randomized, Double-masked Phase 3a Study to Assess Safety and Efficacy of Brolucizumab 6 mg q4 Weeks Compared to Aflibercept 2 mg q4 Weeks in Patients With Neovascular Age-related Macular Degeneration (nAMD) With Persistent Retinal Fluid (MERLIN)
Brief Title: Study of Safety and Efficacy of Brolucizumab 6 mg Dosed Every 4 Weeks Compared to Aflibercept 2 mg Dosed Every 4 Weeks in Patients With Retinal Fluid Despite Frequent Anti-VEGF Injections
Acronym: MERLIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRTH258AUS04
Record Dates: First submitted 2018-10-16; First posted 2018-10-18 (Actual); Results first posted 2022-07-22 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Age-Related Macular Degeneration
Keywords: neovascular age-related macular degeneration; nAMD; intravitreal injection; IVT; anti-VEGF; brolucizumab; aflibercept; EYLEA; double-masked; MERLIN; BEOVU
MeSH Terms: conditions — Macular Degeneration; Neurofibromatosis 2 | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-masked
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brolucizumab (Experimental): Brolucizumab 6 mg dosed every 4 weeks was administered via intravitreal injection for 100 weeks.
  Interventions: Biological: Brolucizumab
- Aflibercept (Active Comparator): Aflibercept 2 mg dosed every 4 weeks was administered via intravitreal injection for 100 weeks.
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Biological: Brolucizumab — 6 mg/0.05mL solution for intravitreal injection
  Other Names: RTH258
  Arms: Brolucizumab
Biological: Aflibercept — 2 mg/0.05mL solution for intravitreal injection
  Other Names: EYLEA
  Arms: Aflibercept

SUMMARY:
This clinical study was designed to compare the safety and efficacy of brolucizumab 6 mg dosed every 4 weeks to aflibercept 2 mg dosed every 4 weeks in those neovascular age-related macular degeneration (nAMD) patients with retinal fluid despite frequent anti-Vascular Endothelial Growth Factor (VEGF) injections.

DETAILED DESCRIPTION:
This was a Phase III, multi-center, randomized, double-masked, parallel group study with 2 masked arms in which participants were randomized 2:1 to receive brolucizumab or aflibercept. All participants had study visits every 4 weeks through week 104.

The study consisted of three study periods:

Screening Period: The screening period lasted up to 2 weeks prior to administration of the first dose of study treatment, dependent upon confirmation of the patient meeting eligibility criteria.

Double-Masked Treatment Period: Participants meeting eligibility criteria entered the treatment period and were randomized in a 2:1 ratio into one of the following 2 masked treatment arms at the Baseline visit: Brolucizumab 6 mg injected every 4 weeks or Aflibercept 2 mg injected every 4 weeks. Treatment period lasted up to week 100.

Safety Follow up Period: Participants were followed up for safety during 4 weeks after the last dose of study treatment. Including the Screening Period, the total study duration for a participant was up to 106 weeks.

Some participants were eligible to continue into an extension study in order to receive treatment with brolucizumab (a) after completing the 104 -week double-masked treatment period, (b) upon meeting all inclusion/exclusion criteria for the extension study, and (c) based on Investigator's judgment that the participant was expected to benefit from treatment with brolucizumab.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of wet age-related macular degeneration (AMD)
* Currently receiving anti-VEGF injections

Exclusion Criteria:

* Active infection or inflammation in either eye
* Significant fibrosis in the study eye
* Recent ocular surgery
* Uncontrolled glaucoma
* Use of medications as specified in the protocol
* Pregnant, nursing
* Of child-bearing potential unless using highly effective method of contraception

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (54):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Oxnard, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, Redlands, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigative Site, Deerfield Beach, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Mt. Dora, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Stuart, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, ‘Aiea, Hawaii
  - Novartis Investigative Site, Wheaton, Illinois
  - Novartis Investigative Site, West Des Moines, Iowa
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, West Monroe, Louisiana
  - Novartis Investigative Site, Waldorf, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Bloomfield, New Jersey
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Fairfield, Ohio
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Abilene, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Harlingen, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Fairfax, Virginia
  - Novartis Investigative Site, Spokane, Washington
- Novartis Investigative Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1133

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brolucizumab | Aflibercept
Started (All randomized Participants) | 356 | 179
Completed | 172 | 86
Not Completed | 184 | 93
Not completed — Study Terminated by Sponsor | 104 | 55
Not completed — Withdrawal by Subject | 57 | 25
Not completed — Death | 10 | 4
Not completed — Lost to Follow-up | 5 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab | Aflibercept | Total
Number analyzed (Participants) | 356 | 179 | 535
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.4 (7.47) | 76.1 (7.80) | 76.3 (7.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 107 | 302
  Male | 161 | 72 | 233
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 347 | 176 | 523
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-Corrected Visual Acuity (BCVA) at Week 52
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. A positive change from baseline represents better functioning.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment. Last observation carried forward (LOCF) was used for the imputation of missing values.
Time Frame: Baseline, week 52
Population: All randomized participants
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Score on a scale | 0.3 (9.02) | 0.9 (6.51)
Statistical Analysis 1: Comparison: Brolucizumab vs Aflibercept; Test type: Superiority; p = 0.4537, Pairwise ANOVA; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-2.1 to 0.9], Standard Error of Mean 0.76

2. Secondary Outcome: Stable Visual Acuity (VA) or Improvement in VA at Week 52 and Week 104
Description: Visual Acuity (VA) was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. VA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of participants with no change or gain in VA compared to baseline was reported. VA stabilization or improvement is defined as a change from baseline no worse than 5 letters loss in VA compared to Baseline.
  Baseline VA was defined as the last measurement on or prior to the baseline visit. VA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: Baseline, weeks 52 and 104
Population: The overall number of participants analyzed includes all randomized participants. The number analyzed per row represents participants with data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 52 | 232 | 132
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 122 | 63

3. Secondary Outcome: Loss in Best-Corrected Visual Acuity (BCVA) of 5 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with loss in BCVA of 5 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: Baseline, weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 31 | 16
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 38 | 17
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 33 | 22
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 34 | 19
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 47 | 15
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 40 | 20
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 46 | 24
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 45 | 24
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 44 | 24
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 46 | 17
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 45 | 17
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 46 | 23
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 50 | 24
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 46 | 17
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 51 | 23
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 47 | 26
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 50 | 28
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 59 | 25
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 48 | 31
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 49 | 27
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 51 | 27
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 37 | 24
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 43 | 24
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 42 | 19
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 40 | 19
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 40 | 23

4. Secondary Outcome: Loss in Best-Corrected Visual Acuity (BCVA) of 10 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with loss in BCVA of 10 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 4 | 6
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 5 | 5
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 9 | 5
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 13 | 4
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 14 | 5
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 8 | 6
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 14 | 9
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 10 | 8
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 9 | 10
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 13 | 5
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 17 | 6
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 20 | 9
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 24 | 7
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 20 | 5
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 21 | 8
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 24 | 10
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 20 | 10
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 21 | 11
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 24 | 13
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 26 | 13
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 20 | 10
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 21 | 14
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 20 | 9
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 18 | 8
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 15 | 7
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 17 | 7

5. Secondary Outcome: Loss in Best-Corrected Visual Acuity (BCVA) of 15 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with loss in BCVA of 15 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 2 | 1
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 2 | 1
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 3 | 2
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 4 | 1
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 5 | 1
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 3 | 1
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 4 | 3
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 6 | 3
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 3 | 4
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 5 | 3
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 6 | 3
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 10 | 3
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 14 | 2
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 13 | 2
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 13 | 3
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 10 | 4
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 10 | 4
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 10 | 3
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 13 | 4
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 12 | 4
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 7 | 6
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 10 | 5
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 11 | 4
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 9 | 4
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 7 | 5
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 10 | 4

6. Secondary Outcome: Gain in Best-Corrected Visual Acuity (BCVA) of 5 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with gain in BCVA of 5 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 94 | 35
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 98 | 43
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 113 | 48
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 119 | 53
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 123 | 47
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 125 | 57
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 129 | 61
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 122 | 57
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 108 | 58
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 111 | 62
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 103 | 50
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 117 | 54
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 108 | 52
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 103 | 48
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 108 | 46
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 106 | 51
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 96 | 46
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 108 | 46
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 107 | 48
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 106 | 50
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 102 | 43
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 93 | 42
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 79 | 36
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 76 | 31
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 70 | 24
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 65 | 28

7. Secondary Outcome: Gain in Best-Corrected Visual Acuity (BCVA) of 10 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with gain in BCVA of 10 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 48 | 18
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 49 | 20
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 62 | 20
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 64 | 28
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 67 | 26
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 77 | 34
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 78 | 36
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 75 | 38
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 69 | 38
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 65 | 37
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 60 | 31
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 66 | 34
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 67 | 32
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 71 | 31
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 67 | 26
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 72 | 28
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 61 | 31
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 62 | 29
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 62 | 24
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 66 | 29
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 59 | 29
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 53 | 24
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 46 | 21
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 50 | 18
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 39 | 15
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 42 | 19

8. Secondary Outcome: Gain in Best-Corrected Visual Acuity (BCVA) of 15 Letters or More
Description: BCVA was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing protocol at an initial testing distance of 4 meters. BCVA min and max possible scores are 0-100 respectively and a higher score represents better functioning. The number of subjects with gain in BCVA of 15 letters or more from baseline was reported for each post-baseline visit.
  Baseline BCVA was defined as the last measurement on or prior to the baseline visit. BCVA assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 353 | 176
  Week 4 | 43 | 14
  Week 8: number analyzed (Participants) | 347 | 174
  Week 8 | 37 | 16
  Week 12: number analyzed (Participants) | 343 | 176
  Week 12 | 51 | 16
  Week 16: number analyzed (Participants) | 341 | 173
  Week 16 | 56 | 23
  Week 20: number analyzed (Participants) | 340 | 171
  Week 20 | 51 | 15
  Week 24: number analyzed (Participants) | 324 | 168
  Week 24 | 64 | 25
  Week 28: number analyzed (Participants) | 327 | 174
  Week 28 | 63 | 28
  Week 32: number analyzed (Participants) | 317 | 166
  Week 32 | 57 | 25
  Week 36: number analyzed (Participants) | 308 | 166
  Week 36 | 50 | 26
  Week 40: number analyzed (Participants) | 299 | 165
  Week 40 | 54 | 26
  Week 44: number analyzed (Participants) | 293 | 157
  Week 44 | 47 | 27
  Week 48: number analyzed (Participants) | 289 | 153
  Week 48 | 50 | 22
  Week 52: number analyzed (Participants) | 282 | 156
  Week 52 | 50 | 27
  Week 56: number analyzed (Participants) | 263 | 139
  Week 56 | 56 | 22
  Week 60: number analyzed (Participants) | 267 | 141
  Week 60 | 56 | 21
  Week 64: number analyzed (Participants) | 266 | 142
  Week 64 | 58 | 22
  Week 68: number analyzed (Participants) | 262 | 139
  Week 68 | 50 | 23
  Week 72: number analyzed (Participants) | 255 | 141
  Week 72 | 49 | 19
  Week 76: number analyzed (Participants) | 260 | 138
  Week 76 | 54 | 14
  Week 80: number analyzed (Participants) | 249 | 136
  Week 80 | 53 | 20
  Week 84: number analyzed (Participants) | 243 | 129
  Week 84 | 44 | 18
  Week 88: number analyzed (Participants) | 225 | 124
  Week 88 | 46 | 18
  Week 92: number analyzed (Participants) | 211 | 112
  Week 92 | 42 | 14
  Week 96: number analyzed (Participants) | 198 | 101
  Week 96 | 39 | 11
  Week 100: number analyzed (Participants) | 174 | 91
  Week 100 | 30 | 11
  Week 104: number analyzed (Participants) | 162 | 86
  Week 104 | 30 | 14

9. Secondary Outcome: Change in Central Subfield Thickness (CST) From Baseline
Description: CST was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. A negative change from baseline is a favorable outcome. CST assessments after start of alternative anti-VEGF treatment in the study eye were censored and imputed by the last value prior to start of alternative treatment. These results were based on analysis using the Last observation carried forward (LOCF) approach for replacement/imputation of censored/missing values and observed data.
Time Frame: as for outcome 3
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: µm
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 178
µm
  Week 4 | -55.1 (2.93) | -29.8 (4.15)
  Week 8 | -59.7 (3.16) | -35.4 (4.48)
  Week 12 | -62.3 (3.24) | -37.3 (4.59)
  Week 16 | -61.7 (3.36) | -39.2 (4.75)
  Week 20 | -64.6 (3.46) | -41.4 (4.90)
  Week 24 | -63.8 (3.61) | -40.8 (5.11)
  Week 28 | -64.3 (3.57) | -35.5 (5.05)
  Week 32 | -65.2 (3.70) | -40.4 (5.23)
  Week 36 | -64.0 (3.81) | -42.3 (5.39)
  Week 40 | -64.9 (3.76) | -38.2 (5.32)
  Week 44 | -66.7 (3.71) | -40.2 (5.24)
  Week 48 | -68.9 (3.76) | -40.7 (5.32)
  Week 52 | -69.0 (3.88) | -37.0 (5.50)
  Week 56 | -70.5 (3.85) | -43.9 (5.45)
  Week 60 | -70.0 (4.00) | -43.6 (5.66)
  Week 64 | -71.2 (3.99) | -41.5 (5.65)
  Week 68 | -71.3 (4.07) | -40.8 (5.77)
  Week 72 | -71.2 (4.08) | -42.6 (5.78)
  Week 76 | -71.4 (4.06) | -46.2 (5.76)
  Week 80 | -72.0 (4.13) | -45.3 (5.85)
  Week 84 | -71.3 (4.15) | -48.4 (5.88)
  Week 88 | -70.9 (4.14) | -44.6 (5.87)
  Week 92 | -69.1 (4.21) | -46.4 (5.97)
  Week 96 | -70.5 (4.13) | -43.5 (5.85)
  Week 100 | -69.8 (4.14) | -47.0 (5.87)
  Week 104 | -71.3 (4.16) | -48.3 (5.90)

10. Secondary Outcome: Number of Participants With Intraretinal Fluid (IRF)
Description: IRF was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. The number of participants with presence of IRF was reported for each post-baseline visit. These results were based on analysis using the Last observation carried forward (LOCF) approach for replacement/imputation of censored/missing values and observed data.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: The overall number of participants analyzed includes all randomized participants. The number analyzed per row represents participants with evaluable data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 349 | 175
  Week 4 | 272 | 132
  Week 8: number analyzed (Participants) | 354 | 178
  Week 8 | 276 | 131
  Week 12: number analyzed (Participants) | 354 | 178
  Week 12 | 279 | 125
  Week 16: number analyzed (Participants) | 354 | 178
  Week 16 | 274 | 126
  Week 20: number analyzed (Participants) | 354 | 178
  Week 20 | 266 | 124
  Week 24: number analyzed (Participants) | 354 | 178
  Week 24 | 266 | 126
  Week 28: number analyzed (Participants) | 354 | 178
  Week 28 | 266 | 128
  Week 32: number analyzed (Participants) | 354 | 178
  Week 32 | 262 | 124
  Week 36: number analyzed (Participants) | 354 | 178
  Week 36 | 255 | 124
  Week 40: number analyzed (Participants) | 354 | 178
  Week 40 | 255 | 121
  Week 44: number analyzed (Participants) | 354 | 178
  Week 44 | 263 | 122
  Week 48: number analyzed (Participants) | 354 | 178
  Week 48 | 265 | 117
  Week 52: number analyzed (Participants) | 355 | 178
  Week 52 | 265 | 120
  Week 56: number analyzed (Participants) | 355 | 178
  Week 56 | 268 | 125
  Week 60: number analyzed (Participants) | 355 | 178
  Week 60 | 278 | 125
  Week 64: number analyzed (Participants) | 355 | 178
  Week 64 | 276 | 126
  Week 68: number analyzed (Participants) | 355 | 178
  Week 68 | 269 | 127
  Week 72: number analyzed (Participants) | 355 | 178
  Week 72 | 271 | 123
  Week 76: number analyzed (Participants) | 355 | 178
  Week 76 | 279 | 122
  Week 80: number analyzed (Participants) | 355 | 178
  Week 80 | 280 | 122
  Week 84: number analyzed (Participants) | 355 | 178
  Week 84 | 274 | 124
  Week 88: number analyzed (Participants) | 355 | 178
  Week 88 | 270 | 122
  Week 92: number analyzed (Participants) | 355 | 178
  Week 92 | 273 | 123
  Week 96: number analyzed (Participants) | 355 | 178
  Week 96 | 270 | 123
  Week 100: number analyzed (Participants) | 355 | 178
  Week 100 | 275 | 126
  Week 104: number analyzed (Participants) | 355 | 178
  Week 104 | 273 | 124

11. Secondary Outcome: Number of Participants With Subretinal Fluid (SRF)
Description: SRF was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. The number of participants with presence of SRF was reported for each post-baseline visit. These results were based on analysis using the Last observation carried forward (LOCF) approach for replacement/imputation of censored/missing values and observed data.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 350 | 176
  Week 4 | 161 | 41
  Week 8: number analyzed (Participants) | 354 | 178
  Week 8 | 193 | 47
  Week 12: number analyzed (Participants) | 354 | 178
  Week 12 | 205 | 46
  Week 16: number analyzed (Participants) | 354 | 178
  Week 16 | 209 | 60
  Week 20: number analyzed (Participants) | 354 | 178
  Week 20 | 200 | 53
  Week 24: number analyzed (Participants) | 354 | 178
  Week 24 | 211 | 59
  Week 28: number analyzed (Participants) | 354 | 178
  Week 28 | 207 | 54
  Week 32: number analyzed (Participants) | 354 | 178
  Week 32 | 211 | 55
  Week 36: number analyzed (Participants) | 354 | 178
  Week 36 | 200 | 69
  Week 40: number analyzed (Participants) | 354 | 178
  Week 40 | 211 | 59
  Week 44: number analyzed (Participants) | 354 | 178
  Week 44 | 211 | 58
  Week 48: number analyzed (Participants) | 354 | 178
  Week 48 | 205 | 62
  Week 52: number analyzed (Participants) | 355 | 178
  Week 52 | 203 | 65
  Week 56: number analyzed (Participants) | 355 | 178
  Week 56 | 211 | 65
  Week 60: number analyzed (Participants) | 355 | 178
  Week 60 | 207 | 64
  Week 64: number analyzed (Participants) | 355 | 178
  Week 64 | 213 | 63
  Week 68: number analyzed (Participants) | 355 | 178
  Week 68 | 212 | 64
  Week 72: number analyzed (Participants) | 355 | 178
  Week 72 | 216 | 72
  Week 76: number analyzed (Participants) | 355 | 178
  Week 76 | 220 | 67
  Week 80: number analyzed (Participants) | 355 | 178
  Week 80 | 220 | 66
  Week 84: number analyzed (Participants) | 355 | 178
  Week 84 | 228 | 67
  Week 88: number analyzed (Participants) | 355 | 178
  Week 88 | 225 | 73
  Week 92: number analyzed (Participants) | 355 | 178
  Week 92 | 222 | 75
  Week 96: number analyzed (Participants) | 355 | 178
  Week 96 | 224 | 73
  Week 100: number analyzed (Participants) | 355 | 178
  Week 100 | 223 | 74
  Week 104: number analyzed (Participants) | 355 | 178
  Week 104 | 227 | 79

12. Secondary Outcome: Number of Participants With Sub-Retinal Pigment Epithelium (Sub-RPE) Fluid
Description: Sub-RPE fluid was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. The number of participants with presence of sub-RPE fluid in participants with sub-RPE fluid at baseline was reported for each post-baseline visit. These results were based on analysis using the Last observation carried forward (LOCF) approach for replacement/imputation of censored/missing values and observed data.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 350 | 176
  Week 4 | 191 | 89
  Week 8: number analyzed (Participants) | 354 | 178
  Week 8 | 213 | 98
  Week 12: number analyzed (Participants) | 354 | 178
  Week 12 | 223 | 98
  Week 16: number analyzed (Participants) | 354 | 178
  Week 16 | 235 | 105
  Week 20: number analyzed (Participants) | 354 | 178
  Week 20 | 232 | 99
  Week 24: number analyzed (Participants) | 354 | 178
  Week 24 | 231 | 101
  Week 28: number analyzed (Participants) | 354 | 178
  Week 28 | 229 | 95
  Week 32: number analyzed (Participants) | 354 | 178
  Week 32 | 237 | 101
  Week 36: number analyzed (Participants) | 354 | 178
  Week 36 | 227 | 101
  Week 40: number analyzed (Participants) | 354 | 178
  Week 40 | 238 | 101
  Week 44: number analyzed (Participants) | 354 | 178
  Week 44 | 235 | 103
  Week 48: number analyzed (Participants) | 354 | 178
  Week 48 | 228 | 105
  Week 52: number analyzed (Participants) | 355 | 178
  Week 52 | 228 | 113
  Week 56: number analyzed (Participants) | 355 | 178
  Week 56 | 240 | 102
  Week 60: number analyzed (Participants) | 355 | 178
  Week 60 | 238 | 107
  Week 64: number analyzed (Participants) | 355 | 178
  Week 64 | 235 | 99
  Week 68: number analyzed (Participants) | 355 | 178
  Week 68 | 231 | 98
  Week 72: number analyzed (Participants) | 355 | 178
  Week 72 | 236 | 96
  Week 76: number analyzed (Participants) | 355 | 178
  Week 76 | 233 | 96
  Week 80: number analyzed (Participants) | 355 | 178
  Week 80 | 234 | 96
  Week 84: number analyzed (Participants) | 355 | 178
  Week 84 | 233 | 100
  Week 88: number analyzed (Participants) | 355 | 178
  Week 88 | 234 | 97
  Week 92: number analyzed (Participants) | 355 | 178
  Week 92 | 236 | 94
  Week 96: number analyzed (Participants) | 355 | 178
  Week 96 | 237 | 101
  Week 100: number analyzed (Participants) | 355 | 178
  Week 100 | 242 | 104
  Week 104: number analyzed (Participants) | 355 | 178
  Week 104 | 237 | 100

13. Secondary Outcome: Number of Participants With Fluid-free Status (no IRF, SRF or Sub-RPE Fluid)
Description: Intraretinal fluid (IRF), Subretinal fluid (SRF) and Sub-Retinal Pigment Epithelium fluid (sub-RPE) were assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. The number of participants with fluid-free status (simultaneous absence of IRF, SRF, and sub-RPE) was reported for each post-baseline visit. These results were based on analysis using the Last observation carried forward (LOCF) approach for replacement/imputation of censored/missing values and observed data.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Participants
  Week 4: number analyzed (Participants) | 347 | 175
  Week 4 | 82 | 16
  Week 8: number analyzed (Participants) | 354 | 178
  Week 8 | 110 | 24
  Week 12: number analyzed (Participants) | 354 | 178
  Week 12 | 120 | 22
  Week 16: number analyzed (Participants) | 354 | 178
  Week 16 | 126 | 23
  Week 20: number analyzed (Participants) | 354 | 178
  Week 20 | 114 | 20
  Week 24: number analyzed (Participants) | 354 | 178
  Week 24 | 122 | 28
  Week 28: number analyzed (Participants) | 354 | 178
  Week 28 | 124 | 23
  Week 32: number analyzed (Participants) | 354 | 178
  Week 32 | 123 | 24
  Week 36: number analyzed (Participants) | 354 | 178
  Week 36 | 111 | 32
  Week 40: number analyzed (Participants) | 354 | 178
  Week 40 | 117 | 23
  Week 44: number analyzed (Participants) | 354 | 178
  Week 44 | 122 | 25
  Week 48: number analyzed (Participants) | 354 | 178
  Week 48 | 116 | 27
  Week 52: number analyzed (Participants) | 355 | 178
  Week 52 | 107 | 25
  Week 56: number analyzed (Participants) | 355 | 178
  Week 56 | 127 | 28
  Week 60: number analyzed (Participants) | 355 | 178
  Week 60 | 125 | 30
  Week 64: number analyzed (Participants) | 355 | 178
  Week 64 | 129 | 28
  Week 68: number analyzed (Participants) | 355 | 178
  Week 68 | 124 | 28
  Week 72: number analyzed (Participants) | 355 | 178
  Week 72 | 133 | 31
  Week 76: number analyzed (Participants) | 355 | 178
  Week 76 | 133 | 25
  Week 80: number analyzed (Participants) | 355 | 178
  Week 80 | 136 | 26
  Week 84: number analyzed (Participants) | 355 | 178
  Week 84 | 135 | 27
  Week 88: number analyzed (Participants) | 355 | 178
  Week 88 | 130 | 32
  Week 92: number analyzed (Participants) | 355 | 178
  Week 92 | 128 | 31
  Week 96: number analyzed (Participants) | 355 | 178
  Week 96 | 127 | 32
  Week 100: number analyzed (Participants) | 355 | 178
  Week 100 | 130 | 34
  Week 104: number analyzed (Participants) | 355 | 178
  Week 104 | 134 | 38

14. Secondary Outcome: Time to First Dry Retina (no IRF or SRF)
Description: Intraretinal fluid (IRF) and Subretinal fluid (SRF) were assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. A dry retina is defined as no IRF or SRF at the respective visit. Kaplan-Meier method was used for estimate of percentiles with 95% CI based on methodology of Brookmeyer and Crowley. Data was censored at the last time when IRF/SRF assessments for fluid-free retina were available for participants who discontinued on/or prior to the time of the start of alternative anti-VEGF treatment. IRF and SRF assessments on unscheduled visits were considered.
Time Frame: Baseline, Up to Week 104 (assessments every 4 weeks)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Days | 87.0 [63.0 to 117.0] | 646.0 [372.0 to NA] — Not estimable, the percentage of participants achieving the event did not reach the required threshold.

15. Secondary Outcome: Time to Sustained Dry Retina (no IRF or SRF at ≥ 2 Consecutive Visits)
Description: Intraretinal fluid (IRF) and Subretinal fluid (SRF) were assessed using Spectral Domain Optical Coherence Tomography (SD-OCT) images. A sustained dry retina is defined as no IRF or SRF at 2 or more consecutive visits. Kaplan-Meier method was used for estimate of percentiles with 95% CI based on methodology of Brookmeyer and Crowley. Data was censored at the last time when IRF/SRF assessments for fluid-free retina were available for participants who discontinued on/or prior to the time of the start of alternative anti-VEGF treatment. IRF and SRF assessments on unscheduled visits were considered.
Time Frame: Baseline, Up to Week 104 (assessments every 4 weeks)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Brolucizumab | Aflibercept
Number analyzed (Participants) | 356 | 179
Days | 148.0 [108.0 to 203.0] | NA [NA to NA] — Not estimable, the percentage of participants achieving the event did not reach the required threshold.

16. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Negative Status
Description: A blood sample was collected for anti-drug antibody assessment. ADA negative status = ADA negative result at the corresponding study visit. The baseline sample was collected prior to first dose of study treatment and the post-baseline assessments were taken at the scheduled timepoints. A negative Titer was used to assess the ADA status for the brolucizumab arm.
Time Frame: Baseline, weeks 4, 12, 24, 36, 52, 76 and 104
Population: The overall number of participants analyzed includes all randomized participants. The number analyzed per row represents participants with data at each time point. This outcome measure was pre-specified for the brolucizumab arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab
Number analyzed (Participants) | 356
Participants
  Baseline: number analyzed (Participants) | 348
  Baseline | 77
  Week 4: number analyzed (Participants) | 347
  Week 4 | 121
  Week 12: number analyzed (Participants) | 341
  Week 12 | 122
  Week 24: number analyzed (Participants) | 324
  Week 24 | 118
  Week 36: number analyzed (Participants) | 308
  Week 36 | 117
  Week 52: number analyzed (Participants) | 287
  Week 52 | 106
  Week 76: number analyzed (Participants) | 261
  Week 76 | 100
  Week 104: number analyzed (Participants) | 236
  Week 104 | 101

17. Secondary Outcome: Free Brolucizumab Serum Concentration
Description: A blood sample was collected for Free Brolucizumab serum concentration assessment. This outcome measure was pre-specified for the brolucizumab arm only. The baseline sample was collected prior to first dose of study treatment and the post-baseline assessments.
  Values below the limit of quantification (BLQ) (<0.5 ng/mL) were replaced by one half of the LLOQ (0.25 ng/mL) in the calculation of the summary statistics. For the Mean score at each visit, if the calculated value was less than 0.5, then "NA" was displayed instead; meaning that the score is below the limit of quantitation (<0.5 ng/mL).
Time Frame: pre-dose a baseline, weeks 4, 12, 24, 36, 52, 76 and 104
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng / mL
Arm/Group | Brolucizumab
Number analyzed (Participants) | 356
ng / mL
  Baseline: number analyzed (Participants) | 346
  Baseline | NA (NA) — Below the limit of quantitation (<0.5 ng/mL)
  Week 4: number analyzed (Participants) | 347
  Week 4 | 0.69 (2.47)
  Week 12: number analyzed (Participants) | 340
  Week 12 | 0.81 (2.33)
  Week 24: number analyzed (Participants) | 324
  Week 24 | 0.69 (2.10)
  Week 36: number analyzed (Participants) | 308
  Week 36 | 0.54 (1.32)
  Week 52: number analyzed (Participants) | 287
  Week 52 | NA (NA) — Below the limit of quantitation (<0.5 ng/mL)
  Week 76: number analyzed (Participants) | 261
  Week 76 | NA (NA) — Below the limit of quantitation (<0.5 ng/mL)
  Week 104: number analyzed (Participants) | 235
  Week 104 | NA (NA) — Below the limit of quantitation (<0.5 ng/mL)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the start of treatment to 4 weeks after end of treatment, assessed up to maximum duration of 104 weeks.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Groups:
- Brolucizumab 6mg: Brolucizumab 6mg
- Aflibercept 2mg: Aflibercept 2mg
- Overall: Overall
Arm/Group | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 10/356 | 4/179 | 14/535
Serious Adverse Events (participants affected / at risk) | 75/356 | 45/179 | 120/535
Other Adverse Events (participants affected / at risk) | 287/356 | 149/179 | 436/535
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=356) | Aflibercept 2mg (N=179) | Overall (N=535)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 4
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 3
Left ventricular failure (Cardiac disorders) | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Angle closure glaucoma - Study eye (Eye disorders) | 1 | 0 | 1
Anterior chamber cell - Study eye (Eye disorders) | 1 | 0 | 1
Anterior chamber flare - Study eye (Eye disorders) | 1 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 0 | 1 | 1
Cataract - Study eye (Eye disorders) | 1 | 1 | 2
Glaucoma - Study eye (Eye disorders) | 1 | 0 | 1
Iridocyclitis - Study eye (Eye disorders) | 1 | 0 | 1
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 1 | 0 | 1
Posterior capsule opacification - Study eye (Eye disorders) | 1 | 0 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 2 | 0 | 2
Retinal haemorrhage - Study eye (Eye disorders) | 1 | 1 | 2
Retinal vasculitis - Study eye (Eye disorders) | 1 | 0 | 1
Retinal vein occlusion - Study eye (Eye disorders) | 1 | 0 | 1
Uveitis - Study eye (Eye disorders) | 4 | 0 | 4
Visual acuity reduced - Study eye (Eye disorders) | 1 | 0 | 1
Vitreal cells - Study eye (Eye disorders) | 1 | 0 | 1
Vitreous haze - Study eye (Eye disorders) | 1 | 0 | 1
Vitritis - Study eye (Eye disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Drowning (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2 | 2
COVID-19 (Infections and infestations) | 2 | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 2 | 1 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 2
Endophthalmitis - Study eye (Infections and infestations) | 1 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 5 | 1 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 2 | 0 | 2
Septic shock (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 1
Corneal abrasion - Study eye (Injury, poisoning and procedural complications) | 1 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Streptococcus test positive - Study eye (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2
Choroid neoplasm - Fellow eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 3
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 2
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 2 | 2 | 4
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 1
Shock (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 6mg (N=356) | Aflibercept 2mg (N=179) | Overall (N=535)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 10
Arrhythmia (Cardiac disorders) | 1 | 2 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 9 | 10 | 19
Tachycardia (Cardiac disorders) | 4 | 0 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 2
Vertigo (Ear and labyrinth disorders) | 8 | 1 | 9
Hypothyroidism (Endocrine disorders) | 5 | 3 | 8
Blepharitis - Fellow eye (Eye disorders) | 10 | 4 | 14
Blepharitis - Study eye (Eye disorders) | 13 | 5 | 18
Cataract - Fellow eye (Eye disorders) | 13 | 3 | 16
Cataract - Study eye (Eye disorders) | 23 | 4 | 27
Cataract nuclear - Fellow eye (Eye disorders) | 4 | 1 | 5
Cataract nuclear - Study eye (Eye disorders) | 8 | 1 | 9
Cataract subcapsular - Study eye (Eye disorders) | 16 | 6 | 22
Chalazion - Study eye (Eye disorders) | 4 | 2 | 6
Conjunctival haemorrhage - Fellow eye (Eye disorders) | 6 | 7 | 13
Conjunctival haemorrhage - Study eye (Eye disorders) | 32 | 14 | 46
Corneal disorder - Study eye (Eye disorders) | 2 | 2 | 4
Corneal oedema - Study eye (Eye disorders) | 3 | 2 | 5
Diabetic retinopathy - Study eye (Eye disorders) | 2 | 2 | 4
Diplopia - Study eye (Eye disorders) | 5 | 1 | 6
Dry age-related macular degeneration - Fellow eye (Eye disorders) | 5 | 0 | 5
Dry age-related macular degeneration - Study eye (Eye disorders) | 10 | 4 | 14
Dry eye - Fellow eye (Eye disorders) | 10 | 3 | 13
Dry eye - Study eye (Eye disorders) | 19 | 4 | 23
Eye irritation - Study eye (Eye disorders) | 4 | 0 | 4
Eye pain - Study eye (Eye disorders) | 9 | 4 | 13
Iridocyclitis - Fellow eye (Eye disorders) | 1 | 2 | 3
Iridocyclitis - Study eye (Eye disorders) | 17 | 3 | 20
Iritis - Study eye (Eye disorders) | 6 | 2 | 8
Lacrimation increased - Study eye (Eye disorders) | 4 | 2 | 6
Meibomian gland dysfunction - Study eye (Eye disorders) | 1 | 2 | 3
Neovascular age-related macular degeneration - Fellow eye (Eye disorders) | 19 | 13 | 32
Neovascular age-related macular degeneration - Study eye (Eye disorders) | 9 | 5 | 14
Ocular hypertension - Fellow eye (Eye disorders) | 1 | 2 | 3
Ocular hypertension - Study eye (Eye disorders) | 3 | 2 | 5
Optic disc haemorrhage - Study eye (Eye disorders) | 2 | 2 | 4
Posterior capsule opacification - Fellow eye (Eye disorders) | 9 | 4 | 13
Posterior capsule opacification - Study eye (Eye disorders) | 8 | 8 | 16
Punctate keratitis - Fellow eye (Eye disorders) | 7 | 2 | 9
Punctate keratitis - Study eye (Eye disorders) | 9 | 5 | 14
Retinal artery embolism - Study eye (Eye disorders) | 4 | 0 | 4
Retinal haemorrhage - Fellow eye (Eye disorders) | 9 | 6 | 15
Retinal haemorrhage - Study eye (Eye disorders) | 16 | 5 | 21
Subretinal fluid - Fellow eye (Eye disorders) | 4 | 2 | 6
Subretinal fluid - Study eye (Eye disorders) | 3 | 2 | 5
Uveitis - Study eye (Eye disorders) | 8 | 3 | 11
Vision blurred - Study eye (Eye disorders) | 7 | 1 | 8
Visual acuity reduced - Fellow eye (Eye disorders) | 4 | 0 | 4
Visual acuity reduced - Study eye (Eye disorders) | 22 | 6 | 28
Vitreal cells - Study eye (Eye disorders) | 3 | 4 | 7
Vitreous detachment - Fellow eye (Eye disorders) | 6 | 3 | 9
Vitreous detachment - Study eye (Eye disorders) | 18 | 5 | 23
Vitreous floaters - Fellow eye (Eye disorders) | 4 | 2 | 6
Vitreous floaters - Study eye (Eye disorders) | 21 | 10 | 31
Vitreous haemorrhage - Study eye (Eye disorders) | 6 | 2 | 8
Vitritis - Study eye (Eye disorders) | 9 | 3 | 12
Constipation (Gastrointestinal disorders) | 3 | 2 | 5
Dental caries (Gastrointestinal disorders) | 9 | 1 | 10
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 4 | 10
Hiatus hernia (Gastrointestinal disorders) | 3 | 3 | 6
Large intestine polyp (Gastrointestinal disorders) | 0 | 3 | 3
Nausea (Gastrointestinal disorders) | 6 | 3 | 9
Toothache (Gastrointestinal disorders) | 2 | 3 | 5
Fatigue (General disorders) | 4 | 0 | 4
Oedema peripheral (General disorders) | 9 | 6 | 15
Drug hypersensitivity (Immune system disorders) | 1 | 2 | 3
Seasonal allergy (Immune system disorders) | 12 | 8 | 20
Bronchitis (Infections and infestations) | 15 | 8 | 23
COVID-19 (Infections and infestations) | 8 | 7 | 15
Cellulitis (Infections and infestations) | 4 | 2 | 6
Chorioretinitis - Study eye (Infections and infestations) | 9 | 1 | 10
Conjunctivitis - Study eye (Infections and infestations) | 4 | 0 | 4
Cystitis (Infections and infestations) | 2 | 3 | 5
Diverticulitis (Infections and infestations) | 2 | 3 | 5
Ear infection (Infections and infestations) | 4 | 3 | 7
Fungal infection (Infections and infestations) | 4 | 3 | 7
Gastroenteritis viral (Infections and infestations) | 2 | 3 | 5
Herpes zoster (Infections and infestations) | 2 | 2 | 4
Hordeolum - Fellow eye (Infections and infestations) | 5 | 3 | 8
Hordeolum - Study eye (Infections and infestations) | 4 | 2 | 6
Influenza (Infections and infestations) | 7 | 2 | 9
Localised infection (Infections and infestations) | 4 | 1 | 5
Nasopharyngitis (Infections and infestations) | 12 | 10 | 22
Pharyngitis (Infections and infestations) | 1 | 2 | 3
Pneumonia (Infections and infestations) | 9 | 1 | 10
Sinusitis (Infections and infestations) | 11 | 11 | 22
Tooth abscess (Infections and infestations) | 4 | 1 | 5
Tooth infection (Infections and infestations) | 4 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 17 | 6 | 23
Urinary tract infection (Infections and infestations) | 36 | 16 | 52
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 4
Bone contusion (Injury, poisoning and procedural complications) | 1 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 23 | 6 | 29
Foreign body in eye - Study eye (Injury, poisoning and procedural complications) | 11 | 2 | 13
Hand fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 3 | 7
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 5 | 1 | 6
Posterior capsule rupture - Study eye (Injury, poisoning and procedural complications) | 0 | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 4 | 1 | 5
Amylase increased (Investigations) | 1 | 3 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2
Blood cholesterol increased (Investigations) | 3 | 4 | 7
Blood creatinine increased (Investigations) | 3 | 2 | 5
Blood glucose increased (Investigations) | 5 | 1 | 6
Blood lactate dehydrogenase increased (Investigations) | 3 | 2 | 5
Blood phosphorus increased (Investigations) | 0 | 2 | 2
Blood potassium increased (Investigations) | 2 | 2 | 4
Blood pressure increased (Investigations) | 6 | 3 | 9
Blood triglycerides increased (Investigations) | 4 | 2 | 6
Blood urea increased (Investigations) | 0 | 2 | 2
Intraocular pressure increased - Fellow eye (Investigations) | 2 | 2 | 4
Intraocular pressure increased - Study eye (Investigations) | 19 | 7 | 26
Lipase increased (Investigations) | 2 | 2 | 4
Mean cell volume increased (Investigations) | 1 | 2 | 3
Monocyte count increased (Investigations) | 2 | 2 | 4
Optic nerve cup/disc ratio increased - Study eye (Investigations) | 0 | 2 | 2
Red blood cell count decreased (Investigations) | 5 | 1 | 6
Urine analysis abnormal (Investigations) | 4 | 2 | 6
White blood cell count increased (Investigations) | 2 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 4 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 1 | 7
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 6 | 21
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 3 | 16
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 3 | 14
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 0 | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 7
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 4
Amnesia (Nervous system disorders) | 2 | 2 | 4
Carotid artery stenosis (Nervous system disorders) | 4 | 1 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 4
Headache (Nervous system disorders) | 6 | 7 | 13
Nerve compression (Nervous system disorders) | 1 | 2 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 4
Sciatica (Nervous system disorders) | 2 | 3 | 5
Anxiety (Psychiatric disorders) | 5 | 4 | 9
Depression (Psychiatric disorders) | 4 | 3 | 7
Insomnia (Psychiatric disorders) | 4 | 1 | 5
Acute kidney injury (Renal and urinary disorders) | 4 | 2 | 6
Haematuria (Renal and urinary disorders) | 7 | 1 | 8
Nephrolithiasis (Renal and urinary disorders) | 3 | 3 | 6
Proteinuria (Renal and urinary disorders) | 12 | 5 | 17
Prostatomegaly (Reproductive system and breast disorders) | 3 | 2 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 6
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Arteriosclerosis (Vascular disorders) | 2 | 3 | 5
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 28 | 23 | 51
Hypotension (Vascular disorders) | 3 | 3 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03710564/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT03710564/SAP_001.pdf